CLINICAL TRIAL: NCT06709508
Title: Retrospective Evaluation of Prosthetic Complications and Peri-implant Bone Resorption in Implant-supported Single Unit Fixed Restorations
Status: Completed | Type: Observational
Sponsor: Özer İşisağ (Other)
Responsible Party: Sponsor-Investigator, Özer İşisağ, Assistant Professor, Afyonkarahisar Health Sciences University
Organization: Afyonkarahisar Health Sciences University (Other)
Other Study IDs: number 2023/4 dated 07.04.2023
Record Dates: First submitted 2024-11-22; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Implant Clinical Survival; Restoration Survival
Keywords: Dental Implant; Implant Supported Fixed Prosthesis; Prosthetic Complication; Bone Loss
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Examination group — This study differs from other clinical studies because the participants of this study consisted of patients undergoing single-member implant-supported restoration treatment at the Department of Prosthodontics, Afyonkarahisar Health Sciences University.

SUMMARY:
This study evaluated the one-year outcomes of implant-supported single-tooth fixed restorations used to replace missing teeth. The aim was to assess the success rates of dental implants and identify potential complications during treatment. A total of 100 individuals aged between 20 and 64 participated in the study. Patients were evaluated one year after their implant treatments through clinical examinations and radiographic imaging.

DETAILED DESCRIPTION:
Aim: The aim of this study was to retrospectively investigate the prosthetic complications and peri-implant bone loss by clinical and radiological examination at the 12th month of implantsupported single-unit fixed restorations.

Materials and Methods: In this retrospective study, 100 volunteer patients, aged between 20 and 64, who received implant-supported single-member fixed restoration treatment, were scanned from the archives and included. The patients were scanned from the archives, called for 12-month follow-ups, and clinical and radiographic evaluations were made. G*Power (G*Power Ver. 3.0.10, Franz Faul, Üniversität Kiel, Germany) package program was used to calculate the sample size. Digital radiographs (periapical-panoramic films) taken from the patients at the end of the implant treatment and at the 12th month follow-up were recorded using Planmeca Romexis® software. ImageJ, a digital image analysis program, was used to evaluate marginal bone loss on radiographs (ImageJ 1.54g- Wayne Rasband and Contributons, National institutes of Health, USA). In evaluating the success and survival of the implants, the criteria in the consensus decisions published at the International Oral Implantology Congress in 2007 were taken as basis. In addition, prosthetic complications such as chipping, screw loosening and decementation; Its relationship with anatomical localization, implant length, implant diameter, abutment type, superstructure material, occlusal table and the condition of the opposing arch was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Participants were required to be over 18
* Not to have any systemic disorders
* Not to smoke
* Have provided consent to the study.

Exclusion Criteria:

* Individuals with any systemic or psychiatric disorders
* Who did not have radiographic data immediately after prosthetic loading

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing single-unit implant-supported restoration treatment at the Department of Prosthodontics, Afyonkarahisar University of Health Sciences
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-04-08 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
Implant survival rate | 12 months
Prosthetic complication rate | 12 months
  This study evaluated the impact of various parameters, including abutment type, occlusal table width, and opposing arch condition, on prosthetic complications such as debonding (descementation), screw loosening, and chipping (porcelain fractures).

CONTACTS AND LOCATIONS:
Locations (1):
- Afyonkarahisar University of Health Sciences Faculty of Dentistry, Department of Prosthodontics, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-07): https://cdn.clinicaltrials.gov/large-docs/08/NCT06709508/Prot_SAP_000.pdf